CLINICAL TRIAL: NCT03243071
Title: Advancing People of Color in Clinical Trials Now: Involvement in Trials Using a Patient-Centered Website: A Community-Engaged Approach
Acronym: ACT Now
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-00170
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Recruitment
Keywords: Medical Care; Racial Discrimination; Poor Health Literacy; Medical Care Disparities
MeSH Terms: conditions — Racism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will have access to culturally tailored website.
  Interventions: Behavioral: Tailored Website
- Control Group (Active Comparator): Participants in the control group will have access to NYU 's standard trial participation website.
  Interventions: Behavioral: Standard Website

INTERVENTIONS:
Behavioral: Tailored Website — Participants randomized to the intervention arm will have free access to a password protected interactive culturally and linguistically tailored website via a tablet device. No private identifiable data about you will be collected. Participants will receive a brief 10-minute tutorial by a trained research assistant on login procedures and use of the website.
  Arms: Intervention Group
Behavioral: Standard Website — Participants randomized to the control condition will have free access to the NYU standard clinical trials website. Participants in the control condition will have access to the tailored website at the date of study completion (no later than 6 months' post-date of enrollment).
  Arms: Control Group

SUMMARY:
The purpose pf this study is to evaluate the comparative effectiveness of a culturally and linguistically tailored clinical trial literacy website in increasing likelihood of participating in clinical trials. To achieve this objective,a randomized group design will address the following patient-centered outcomes: willingness to enroll in clinical trials and behavioral intent as well as likelihood of referring others to enroll in such trials) before and after exposure to a culturally-tailored clinical trial literacy website. Health literacy will be measured both before and post exposure to tailored messages. Participants will be randomized into two groups. The intervention group (n=50) will have access to culturally tailored website. Participants in the control group (n=50) will have access to NYU 's standard trial participation website.

DETAILED DESCRIPTION:
Compelling evidence demonstrates racial/ethnic disparities in health and healthcare in the United States. These disparities arise from various factors including unequal access to adequate medical care, perceived racial discrimination, and poor health literacy.The Center for Healthful Behavior Change (CHBC) has been involved in numerous initiatives to eradicate health disparities and have implemented NIH-funded interventions to address inequities in health. Interventions targeting patient-centered outcomes have been suboptimal because of inadequate infrastructure to support equitable contributions from stakeholders (patients, providers, and community leaders) in all aspects of the research process. This is crucial to promote sustainable effects regarding minority patients' ability to make informed decisions about participating in existing clinical trials. This study will address this gap, bringing together academic investigators and important stakeholders to develop a website providing access to culturally tailored videos to enhance awareness of clinical trial, health literacy, thus promoting participation in existing clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported race/ethnicity as African American, African, Caribbean American or black men and women
* accessible by telephone
* no plans to move away from the region within the year following enrollment; consent to participate.

Exclusion Criteria:

* Progressive medical illness in which disability or death is expected within one year
* impaired cognitive or functional ability, which would preclude meaningful participation in the study
* stated intention to move within the same year of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Girardin Jean-Louis, Ph.D., Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chung A, Seixas A, Williams N, Senathirajah Y, Robbins R, Newsome Garcia V, Ravenell J, Jean-Louis G. Development of "Advancing People of Color in Clinical Trials Now!": Web-Based Randomized Controlled Trial Protocol. JMIR Res Protoc. 2020 Jul 14;9(7):e17589. doi: 10.2196/17589. PMID 32673274

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 59 | 53
Completed | 59 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: The intervention group (n=50) will have access to culturally tailored website.
  Tailored Website: Participants randomized to the intervention arm will have free access to a password protected interactive culturally and linguistically tailored website via a tablet device. No private identifiable data about you will be collected. Participants will receive a brief 10-minute tutorial by a trained research assistant on login procedures and use of the website.
- Control Group: Participants in the control group (n=50) will have access to NYU 's standard trial participation website.
  Standard Website: Participants randomized to the control condition will have free access to the NYU standard clinical trials website. Participants in the control condition will have access to the tailored website at the date of study completion (no later than 6 months' post-date of enrollment).
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 59 | 53 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (15.98) | 43 (15.03) | 43 (15.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 27 | 73
  Male | 13 | 26 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 7 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 36 | 83
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 59 | 53 | 112

OUTCOME MEASURES:

1. Primary Outcome: ACTNOW! Clinical Trial Knowledge Assessment Score
Description: 26 statements involved in assessing the participants' knowledge of clinical trials. The total range of score is 0-104; the higher the score, the higher the level of knowledge.
Time Frame: Baseline
Population: The discrepancy in overall number of participants analyzed with numbers provided in the participant flow module lies with over enrollment of study subjects to account for attrition loss and analysis only being done for those participants who had complete data.
  The two arms (intervention and control groups) are further divided into pairs for statistical analysis purposes (paired t-tests).
Measure: Mean (Standard Deviation); unit: score
Groups:
- Intervention Group (Pair 1); Intervention Group (Pair 2): The intervention group will have access to culturally tailored website.
  Tailored Website: Participants randomized to the intervention arm will have free access to a password protected interactive culturally and linguistically tailored website via a tablet device. No private identifiable data about you will be collected. Participants will receive a brief 10-minute tutorial by a trained research assistant on login procedures and use of the website.
- Control Group (Pair 3); Control Group (Pair 4): Participants in the control group will have access to NYU 's standard trial participation website.
  Standard Website: Participants randomized to the control condition will have free access to the NYU standard clinical trials website. Participants in the control condition will have access to the tailored website at the date of study completion (no later than 6 months' post-date of enrollment).
Arm/Group | Intervention Group (Pair 1) | Intervention Group (Pair 2) | Control Group (Pair 3) | Control Group (Pair 4)
Number analyzed (Participants) | 47 | 33 | 49 | 25
score | 93.89 (9.98) | 93.58 (9.69) | 94.88 (11.80) | 97.88 (11.45)

2. Primary Outcome: Clinical Trial Knowledge Assessment Score
Description: as for outcome 1
Time Frame: Month 1
Population: The discrepancy in overall number of participants analyzed with numbers provided in the participant flow module lies with over enrollment of study subjects to account for attrition loss and analysis only being done for those participants who had complete data.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention Group (Pair 1) | Control Group (Pair 3)
Number analyzed (Participants) | 47 | 49
score | 101.89 (10.37) | 99.67 (10.94)

3. Primary Outcome: Clinical Trial Knowledge Assessment Score
Description: as for outcome 1
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Intervention Group (Pair 2) | Control Group (Pair 4)
Number analyzed (Participants) | 33 | 25
score | 98.00 (11.99) | 98.32 (8.46)

4. Primary Outcome: ACTNOW! Self-Efficacy Score
Description: A 4-item perceived effectiveness scale was used to assess the perceived persuasiveness of the message. The total range of score is 0-16; the higher the score, the higher the level of self-efficacy.
Time Frame: Baseline
Population: The two arms (intervention and control groups) are further divided into pairs for statistical analysis purposes (paired t-tests).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Group (Pair 3): Participants in the control group (n=50) will have access to NYU 's standard trial participation website.
  Standard Website: Participants randomized to the control condition will have free access to the NYU standard clinical trials website. Participants in the control condition will have access to the tailored website at the date of study completion (no later than 6 months' post-date of enrollment).
Arm/Group | Intervention Group (Pair 1) | Intervention Group (Pair 2) | Control Group (Pair 3) | Control Group (Pair 4)
Number analyzed (Participants) | 47 | 33 | 49 | 25
score on a scale | 10.13 (4.19) | 10.06 (4.49) | 11.16 (3.08) | 11.04 (3.08)

5. Primary Outcome: Self-Efficacy Score
Description: A 4-item perceived effectiveness scale, adapted from Fishbein et al. (2002) was used to assess the perceived persuasiveness of the message. The total range of score is 0-16; the higher the score, the higher the level of self-efficacy.
Time Frame: Month 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group (Pair 1) | Control Group (Pair 3)
Number analyzed (Participants) | 47 | 49
score on a scale | 12.06 (3.35) | 12.02 (3.40)

6. Primary Outcome: Self-Efficacy Score
Description: as for outcome 5
Time Frame: Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group (Pair 2) | Control Group (Pair 4)
Number analyzed (Participants) | 33 | 25
score on a scale | 12.42 (3.40) | 11.88 (3.10)

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/53
Other Adverse Events (participants affected / at risk) | 0/59 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT03243071/Prot_SAP_000.pdf